CLINICAL TRIAL: NCT01292265
Title: A Phase 3b, Open Label, Multicenter, Exploratory Study to Assess Changes in Joint Inflammation Using Ultrasonography in Subjects With Rheumatoid Arthritis Treated for 12 Weeks With Certolizumab Pegol
Brief Title: A 12 Week Study to Assess Changes in Joint Inflammation Using Ultrasonography in Patients With Rheumatoid Arthritis (RA)
Acronym: SWIFT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termination of study due to low enrollment. There were no safety issues.
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA0033
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2012-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis; Joint pain; Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Arthralgia; Inflammation | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CZP 200 mg (Experimental): Certolizumab Pegol (CZP) subcutaneous (sc) injections of 400 mg at Weeks 0, 2 and 4, followed by 200 mg at Weeks 6, 8 and 10.
  Interventions: Biological: Certolizumab Pegol

INTERVENTIONS:
Biological: Certolizumab Pegol — Certolizumab Pegol (CZP) subcutaneous (sc) injections of 400 mg at Weeks 0, 2 and 4, followed by 200 mg at Weeks 6, 8 and 10.
  Other Names: Cimzia; CZP

SUMMARY:
To evaluate the changes in joint inflammation produced by Cimzia over 12 week Treatment period measured by Power/Color Doppler and Gray scale Ultrasound.

DETAILED DESCRIPTION:
Since only 3 subjects were enrolled in this study, the efficacy data is not interpretable and will not be presented. Only Adverse Event (AE) data will be summarized in a table, with frequency counts and percentages.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with adult-onset Rheumatoid Arthritis (RA) >6 months and <3 years
* Active RA
* Must have failed at least one disease modifying Anti Rheumatic Drug (DMARD) treatment
* Subject can have attempted no more than one previous Anti Tumor Necrosis factor (anti-TNF) and discontinued due to drug intolerance

Exclusion Criteria:

* Subject cannot have a second non-inflammatory musculoskeletal condition
* Subject cannot have a diagnosis of any other inflammatory arthritis
* Subject cannot have any previously infected prosthesis
* Subject cannot have arthroplasties in any of the joints assessed in the study
* Subject cannot have a history of chronic infections
* Subject cannot have known Tuberculosis (TB) disease, high risk of acquiring TB, or latent TB infection
* Subject cannot have a history of or current Lymphoproliferative disorder
* Subject cannot have known Human Immunodeficiency Virus (HIV) infection
* Subject cannot have received a live or attenuated vaccine within 8 weeks
* Subject cannot have current or history of malignancy
* Subject cannot have a history of blood disorders
* Subject cannot have a current or recent history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological or cerebral disease
* Subjects must not have a history of adverse reaction to Polyethylene glycol (PEG), a protein medicinal product, or ultrasound gel applied to the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (6):
- United States (6):
  - 10, Los Angeles, California
  - 4, Walnut Creek, California
  - 8, Wheaton, Maryland
  - 1, Voorhees Township, New Jersey
  - 6, Rochester, New York
  - 7, Franklin, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started in February 2011. It was subsequently terminated due to low enrollment.
  Baseline characteristics refer to the Safety Set (SS). The Safety Set (SS) consisted of all patients included in this study receiving treatment with Certolizumab Pegol (CZP) at least once.
  There was a total of 3 subjects enrolled in this study.
Pre-assignment Details: Since only 3 subjects were enrolled in this study, the efficacy data is not interpretable and will not be presented. Only Adverse Event (AE) data will be summarized in a table, with frequency counts and percentages.
Period: Overall Study
Arm/Group | CZP 200 mg
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CZP 200 mg
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Week 0) in the Modified Ultrasound-7 Joint (mUS7) Sumscore at Week 12
Time Frame: From Baseline (Week 0) to Week 12
Population: Since only 3 subjects were enrolled in this study, the efficacy data is not interpretable and will not be presented.
Arm/Group | CZP 200 mg
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline (Week 0) in the Clinical Disease Activity Index (CDAI) at Week 12
Time Frame: From Baseline (Week 0) to Week 12
Population: Since only 3 subjects were enrolled in this study, the efficacy data is not interpretable and will not be presented.
Arm/Group | CZP 200 mg
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline (Week 0) in C-reactive Protein (CRP) at Week 12
Time Frame: From Baseline (Week 0) to Week 12
Population: Since only 3 subjects were enrolled in this study, the efficacy data is not interpretable and will not be presented.
Arm/Group | CZP 200 mg
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline (Week 0) in Erythrocyte Sedimentation Rate (ESR) at Week 12
Time Frame: From Baseline (Week 0) to Week 12
Population: Since only 3 subjects were enrolled in this study, the efficacy data is not interpretable and will not be presented.
Arm/Group | CZP 200 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected during the course of the trial, which was approximately 12 weeks per subject. Since only 3 subjects were enrolled in this study, only AE data will be summarized in a table, with frequency counts and percentages.
Description: Adverse Events refer to the Safety Set (SS). The Safety Set (SS) consisted of all patients included in this study receiving treatment with Certolizumab Pegol (CZP) at least once.
Arm/Group | CZP 200 mg
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CZP 200 mg (N=3)
Nasopharyngitis (Infections and infestations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.